CLINICAL TRIAL: NCT05899881
Title: A Pilot Study Investigating the Effects of a Yoga Intervention on Health and Well-Being Among a Diverse Sample of Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brock University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Kimberley Gammage, Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-205
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Yoga; Body image; Embodiment; Self-objectification; Pilot

STUDY DESIGN:
Intervention Model Description: Pilot study in which participants are randomly assigned to either a yoga group or waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga intervention (Experimental): 10 week yoga intervention; one yoga session per week, 60 minutes in length
  Interventions: Behavioral: Yoga intervention
- Control (No Intervention): Waitlist control asked not to make any lifestyle changes over the 10 week intervention period, and not engage in yoga

INTERVENTIONS:
Behavioral: Yoga intervention — 10 weeks of Hatha yoga, once per week, 60 minutes per class
  Arms: Yoga intervention

SUMMARY:
The goal of this pilot study is to examine how to design a large-scale randomized control trial examining yoga as a way to improve positive body image in men and women across the lifespan. The main questions it will answer are:

* Is the study acceptable to participants?
* Is recruitment, adherence, and retention adequate?
* Are study procedures appropriate?
* What is the preliminary effect of yoga on embodiment (sense of connection with the body), self-objectification (evaluating oneself based on outer appearance rather than internal functions) and body appreciation?

Participants will either take part in a 10-week yoga program or a control condition (where they will be asked to not change their lifestyle). They will complete online questionnaires at the start, middle and end of the 10-weeks.

DETAILED DESCRIPTION:
The purposes of this pilot study are:

* To evaluate the feasibility and acceptability of a randomized control trial by assessing participant retention, data collection procedures, and adherence to engaging in a supervised Hatha yoga intervention (or control group).
* To examine preliminary effects of a yoga intervention on embodiment, self-objectification, and positive body image (i.e., body appreciation) among a diverse sample of adults men and women.

Specifically, we will test whether a 10-week Hatha yoga program will contribute to improvements in body appreciation via a) greater embodiment, and b) lower self-objectification This will allow us to calculate effect sizes for sample size calculations for future randomized controlled trials.

Clearance from the university Research Ethics Board will be obtained prior to study commencement. Participants will be recruited from community centres, social media, and traditional media in the Niagara Region. Potential participants will contact the researcher if they are interested in participating. Eligible and interested participants will be provided with a link to the baseline survey via Qualtrics, where they will complete informed consent, demographic information and measures of physical activity and body image. Once questionnaires have been completed, participants will be randomly assigned (using Microsoft Excel to randomize) to either the yoga or control group. They will be provided with instructions for their group at this time via email. They will then undergo either the 10-week yoga intervention or the control condition (see below for descriptions).

Participants will be asked to complete the same physical activity and body image measures during week 5 and at the end of 10 weeks via Qualtrics. At the final time point, participants will also be asked to complete feasibility measures (e.g., acceptability, appropriateness and feasibility of the intervention and control groups), as well as a series of questions asking about their perceptions of the yoga intervention or control group. Upon completion of all measures, participants will be fully debriefed as to the true purpose of the study and the use of deception (i.e., true purpose of the study related to positive body image); they will then be asked to provide continuing informed consent. In addition, the yoga instructors will also be asked a series of questions regarding their perceptions of the yoga intervention.

Yoga Intervention: Participants randomized to the yoga intervention will be asked to not make changes to other aspects of their lifestyle including their regular physical activity. Instructors are provided with guidelines regarding the format, poses, language, and themes of each class, but within those guidelines, instructors can design their own class each week. Each week, there will be a theme promoting empowerment or positive body image; instructors will be asked to choose specific poses, mantras, mudras, and affirmations to reinforce the theme of that week. Modifications to poses will be provided by the instructor. Yoga equipment will be provided during each yoga session.

Each yoga class will be audio recorded to document the content of the yoga classes to ensure guidelines for the classes are followed. Attendance will be recorded at each class to track adherence.

Instructors: The instructors will have a minimum of two years of teaching experience with diverse populations and must be a registered yoga teacher (e.g., RYT200/CYA-RYT200), meaning they have completed a minimum of 200 hours of yoga teacher training in a Yoga Alliance Foundation/Canadian Yoga Alliance recognized teacher training. Clothing will be standardized across instructors and appropriate for Hatha Yoga (e.g., yoga pants and a t-shirt or tank top). Instructors will be provided with an instructor manual that outlines the basic class structure and poses, themes, and language. The instructor will be blinded to the true study purpose. Instructors will then be asked to create a sample class, following the manual guidelines to teach a practice class to the research team for feedback.

Language and Themes Used in a Hatha Yoga Class

Control group: Participants randomized to the control group will be asked not to practice yoga for the duration of the study. Participants will be informed that they can engage in their regular physical activity routines and not change any other lifestyle factors. Participants in the control group will be offered one free yoga class in-person at the end of the study and offered one free pre-recorded video of a yoga class (from the intervention) at the end of the study.

Participants: A target of approximately 65 adults will be recruited (based on expected dropout of 30%).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Able to read and understand English.
* Community-dwelling and residing in Niagara Region.
* Can attend sessions at the Brock Functional Inclusive Training Centre (Bfit).
* Have not participated in yoga in the past 12 months.
* Must have no underlying medical conditions that would prevent them from practicing Hatha Yoga.

Exclusion Criteria:

* Unable to provide clearance for physical activity as assessed by Get Active questionnaire (CSEP and Health Canada, www.csep.ca) or doctor's note
* Average score >4 on the Body Appreciation Scale-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Body appreciation | Baseline
  Body Appreciation Scale-2 (Tylka & Wood-Barcalow, 2015); 10 items, with each one rated on a 5-point scale ranging from 1 = never to 5 = always. Scores on the BAS-2 are averaged where higher scores represent higher levels of body appreciation.
Body appreciation | 5 weeks
  Body Appreciation Scale-2 (Tylka & Wood-Barcalow, 2015); 10 items, with each one rated on a 5-point scale ranging from 1 = never to 5 = always. Scores on the BAS-2 are averaged where higher scores represent higher levels of body appreciation.
Body appreciation | 10 weeks
  Body Appreciation Scale-2 (Tylka & Wood-Barcalow, 2015); 10 items, with each one rated on a 5-point scale ranging from 1 = never to 5 = always. Scores on the BAS-2 are averaged where higher scores represent higher levels of body appreciation.

SECONDARY OUTCOMES:
Embodiment | Baseline
  Body Responsiveness Scale (Daubenmier, 2005); Each item is rated on a 7-point scale from 1 = not at all true of me to 7 = always true of me. Higher scores indicate greater body responsiveness.
Embodiment | 5 weeks
  Body Responsiveness Scale (Daubenmier, 2005); Each item is rated on a 7-point scale from 1 = not at all true of me to 7 = always true of me. Higher scores indicate greater body responsiveness.
Embodiment | 10 weeks
  Body Responsiveness Scale (Daubenmier, 2005); Each item is rated on a 7-point scale from 1 = not at all true of me to 7 = always true of me. Higher scores indicate greater body responsiveness.
Self-objectification | Baseline
  Self-Objectification Beliefs and Behaviours Scale (Lindner & Tantleff-Dunn, 2017); 14 items, ranging from 1= strongly disagree to 5= strongly agree. Higher scores indicate higher levels of self-objectification.
Self-objectification | 5 weeks
  Self-Objectification Beliefs and Behaviours Scale (Lindner & Tantleff-Dunn, 2017); 14 items, ranging from 1= strongly disagree to 5= strongly agree. Higher scores indicate higher levels of self-objectification.
Self-objectification | 10 weeks
  Self-Objectification Beliefs and Behaviours Scale (Lindner & Tantleff-Dunn, 2017); 14 items, ranging from 1= strongly disagree to 5= strongly agree. Higher scores indicate higher levels of self-objectification.
Body surveillance | Baseline
  Objectified Body Consciousness Scale (McKinley & Hyde, 1996); 7 items rated on 7-point scale ranging from 1 = strongly disagree to 7 = strongly agree; higher scores represent higher survellance
Body surveillance | 5 weeks
  Objectified Body Consciousness Scale (McKinley & Hyde, 1996); 7 items rated on 7-point scale ranging from 1 = strongly disagree to 7 = strongly agree; higher scores represent higher survellance
Body surveillance | 10 weeks
  Objectified Body Consciousness Scale (McKinley & Hyde, 1996); 7 items rated on 7-point scale ranging from 1 = strongly disagree to 7 = strongly agree; higher scores represent higher survellance
Functionality appreciation | Baseline
  Functional Appreciation Scale (Alleva et al., 2017); seven items, each one rated from 1= strongly disagree to 5 = strongly agree. Scores on the FAS are averaged where higher scores indicate higher levels of functionality appreciation.
Functionality appreciation | 5 weeks
  Functional Appreciation Scale (Alleva et al., 2017); seven items, each one rated from 1= strongly disagree to 5 = strongly agree. Scores on the FAS are averaged where higher scores indicate higher levels of functionality appreciation.
Functionality appreciation | 10 weeks
  Functional Appreciation Scale (Alleva et al., 2017); seven items, each one rated from 1= strongly disagree to 5 = strongly agree. Scores on the FAS are averaged where higher scores indicate higher levels of functionality appreciation.
Authentic body pride | Baseline
  Body Self-Conscious Emotions Scale (Castonguay et al., 2014) - Authentic pride subscale - 4 items rated on a 7-point Likert scale from 1 = not at all true of me to 7 = very true of me). Higher scores indicate greater amounts of each emotion.
Authentic body pride | 5 weeks
  Body Self-Conscious Emotions Scale (Castonguay et al., 2014) - Authentic pride subscale - 4 items rated on a 7-point Likert scale from 1 = not at all true of me to 7 = very true of me). Higher scores indicate greater amounts of each emotion.
Authentic body pride | 10 weeks
  Body Self-Conscious Emotions Scale (Castonguay et al., 2014) - Authentic pride subscale - 4 items rated on a 7-point Likert scale from 1 = not at all true of me to 7 = very true of me). Higher scores indicate greater amounts of each emotion.
Fitness-related authentic body pride | Baseline
  Body Self-Conscious Emotions - Fitness Related Instrument (Castonguay et al., 2016) - Authentic body pride - Participants rate the degree to which 4 statements apply to them on a 5-point Likert scale from 1 = never to 5 = always. Higher scores indicate higher levels of fitness aspects of authentic pride.
Fitness-related authentic body pride | 5 weeks
  Body Self-Conscious Emotions - Fitness Related Instrument (Castonguay et al., 2016) - Authentic body pride - Participants rate the degree to which 4 statements apply to them on a 5-point Likert scale from 1 = never to 5 = always. Higher scores indicate higher levels of fitness aspects of authentic pride.
Fitness-related authentic body pride | 10 weeks
  Body Self-Conscious Emotions - Fitness Related Instrument (Castonguay et al., 2016) - Authentic body pride - Participants rate the degree to which 4 statements apply to them on a 5-point Likert scale from 1 = never to 5 = always. Higher scores indicate higher levels of fitness aspects of authentic pride.
Body image flexibility | Baseline
  Body Image-Acceptance and Action Questionnaire (Sandoz et al., 2013); Participants rate the degree to which each of 12 statement applies to them on a 7-point Likert scale from 1 = never true to 7 = always true. Higher scores indicate higher levels of body image flexibility
Body image flexibility | 5 weeks
  Body Image-Acceptance and Action Questionnaire (Sandoz et al., 2013); Participants rate the degree to which each of 12 statement applies to them on a 7-point Likert scale from 1 = never true to 7 = always true. Higher scores indicate higher levels of body image flexibility
Body image flexibility | 10 weeks
  Body Image-Acceptance and Action Questionnaire (Sandoz et al., 2013); Participants rate the degree to which each of 12 statement applies to them on a 7-point Likert scale from 1 = never true to 7 = always true. Higher scores indicate higher levels of body image flexibility
Satisfaction with function of the body and appearance of the body as assessed by Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); | Baseline
  Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); Participants rate the degree to which each of 9 statements is true of them on a 7-point Likert scale from 1 = very dissatisfied to 7 = very satisfied. Higher scores indicated higher levels of body satisfaction.
Satisfaction with function of the body and appearance of the body as assessed by Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); | 5 weeks
  Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); Participants rate the degree to which each of 9 statements is true of them on a 7-point Likert scale from 1 = very dissatisfied to 7 = very satisfied. Higher scores indicated higher levels of body satisfaction.
Satisfaction with function of the body and appearance of the body as assessed by Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); | 10 weeks
  Satisfaction with Body Function and Body Appearance Scale (Reboussin et al., 2000); Participants rate the degree to which each of 9 statements is true of them on a 7-point Likert scale from 1 = very dissatisfied to 7 = very satisfied. Higher scores indicated higher levels of body satisfaction.
Attendance | 10 weeks
  Number of sessions out of 10 attended
Adherence | 10 weeks
  Proportion of total sessions attended by participants
Drop-out | Baseline
  Number and percent of participants lost
Drop-out | 5 weeks
  Number and percent of participants lost
Drop-out | 10 weeks
  Number and percent of participants lost
Retention | Baseline
  Proportion of participants from each group with complete data on each outcome measure
Retention | 5 weeks
  Proportion of participants from each group with complete data on each outcome measure
Retention | 10 weeks
  Proportion of participants from each group with complete data on each outcome measure
Acceptability of the Intervention as assessed by Weiner et al.'s (2017) acceptability measure | 10 weeks
  Acceptability of Intervention Measure (adapted from Weiner et al., 2017); comprised of 5 items; each item rated on a 5-point scale ranging from 1 = completely disagree to 5 = completely agree. Assesses perception among participants that the yoga intervention is agreeable, palatable, or satisfactory. Higher scores represent higher acceptability
Feasibility of intervention as assessed by Weiner et al.'s (2017) feasibility measure | 10 weeks
  Feasibility of Intervention Measure (adapted from Weiner et al., 2017); 5-item measure, with each item rated on a 5-point scale ranging from 1 = completely disagree to 5 = completely agree. Assesses the extent to which the yoga intervention can be successfully carried out in this setting.Higher scores represent higher feasibility
Appropriateness of intervention as assessed by Weiner et al.'s (2017) appropriateness measure | 10 weeks
  Intervention Appropriateness Measure (adapted from Weiner et al., 2017); 5-item measure, with each item rated on a 5-point scale ranging from 1 = completely disagree to 5 = completely agree. Assesses perceived fit, relevance, or compatibility of the yoga intervention in this setting and sample. Higher scores represent higher appropriateness
Interest in engaging in the yoga intervention | Baseline
  Number of participants (by age and gender) who express interest in the study by contacting the research team
Recruitment | Baseline
  Number and percent of men and women, age group, and weight status group enrolled

OTHER OUTCOMES:
Physical activity | Baseline
  Godin Leisure Time Physical Activity Questionnaire (Godin & Shephard, 1985); Participants are asked to report the number of times they engaged in mild, moderate, and strenuous physical activity for greater than 15 min during the last 7-day period. A total score is calculated by multiplying the frequencies of mild, moderate, and strenuous activity by corresponding metabolic equivalent task values (three, five, and nine, respectively) and summing the scores. Higher scores are reflective of greater energy expenditure.
Physical activity | 5 weeks
  Godin Leisure Time Physical Activity Questionnaire (Godin & Shephard, 1985); Participants are asked to report the number of times they engaged in mild, moderate, and strenuous physical activity for greater than 15 min during the last 7-day period. A total score is calculated by multiplying the frequencies of mild, moderate, and strenuous activity by corresponding metabolic equivalent task values (three, five, and nine, respectively) and summing the scores. Higher scores are reflective of greater energy expenditure.
Physical activity | 10 weeks
  Godin Leisure Time Physical Activity Questionnaire (Godin & Shephard, 1985); Participants are asked to report the number of times they engaged in mild, moderate, and strenuous physical activity for greater than 15 min during the last 7-day period. A total score is calculated by multiplying the frequencies of mild, moderate, and strenuous activity by corresponding metabolic equivalent task values (three, five, and nine, respectively) and summing the scores. Higher scores are reflective of greater energy expenditure.
Stress | Baseline
  Perceived Stress Scale (Cohen et al., 1983). 10 items rated on a 5-point Likert scale from 0 = never to 4 = very often. Higher scores indicate higher levels of perceived stress.
Stress | 5 weeks
  Perceived Stress Scale (Cohen et al., 1983). 10 items rated on a 5-point Likert scale from 0 = never to 4 = very often. Higher scores indicate higher levels of perceived stress.
Stress | 10 weeks
  Perceived Stress Scale (Cohen et al., 1983). 10 items rated on a 5-point Likert scale from 0 = never to 4 = very often. Higher scores indicate higher levels of perceived stress.
Depression | Baseline
  Center for Epidemiologic Studies Depression Scale (Radloff, 1997); Participants rate the degree to which each statement is true of them on a range from 0 = rarely or none to 3 = most or almost all the time. Questions scores are then summed to provide an overall score ranging from 0 to 60. Higher scores indicate greater depression symptoms.
Depression | 5 weeks
  Center for Epidemiologic Studies Depression Scale (Radloff, 1997); Participants rate the degree to which each statement is true of them on a range from 0 = rarely or none to 3 = most or almost all the time. Questions scores are then summed to provide an overall score ranging from 0 to 60. Higher scores indicate greater depression symptoms.
Depression | 10 weeks
  Center for Epidemiologic Studies Depression Scale (Radloff, 1997); Participants rate the degree to which each statement is true of them on a range from 0 = rarely or none to 3 = most or almost all the time. Questions scores are then summed to provide an overall score ranging from 0 to 60. Higher scores indicate greater depression symptoms.
Participant perceptions of intervention | 10 weeks
  Open ended questions
Instructor perceptions | 10 weeks
  Open ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley L Gammage, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University - Brock Functional Inclusive Training Centre, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Tylka TL, Wood-Barcalow NL. What is and what is not positive body image? Conceptual foundations and construct definition. Body Image. 2015 Jun;14:118-29. doi: 10.1016/j.bodyim.2015.04.001. Epub 2015 Apr 25. PMID 25921657
- [Background] Alleva JM, Tylka TL, van Oorsouw K, Montanaro E, Perey I, Bolle C, Boselie J, Peters M, Webb JB. The effects of yoga on functionality appreciation and additional facets of positive body image. Body Image. 2020 Sep;34:184-195. doi: 10.1016/j.bodyim.2020.06.003. Epub 2020 Jul 1. PMID 32622294
- [Background] Alleva JM, Tylka TL, Kroon Van Diest AM. The Functionality Appreciation Scale (FAS): Development and psychometric evaluation in U.S. community women and men. Body Image. 2017 Dec;23:28-44. doi: 10.1016/j.bodyim.2017.07.008. Epub 2017 Aug 17. PMID 28822275
- [Background] Castonguay, A. L., Sabiston, C. M., Kowalski, K. C., & Wilson, P. M. Introducing an instrument to measure body and fitness-related self-conscious emotions: The BSE-FIT. Psychology of Sport and Exercise. 2016; 23: 1-12.
- [Background] Castonguay AL, Pila E, Wrosch C, Sabiston CM. Body-related self-conscious emotions relate to physical activity motivation and behavior in men. Am J Mens Health. 2015 May;9(3):209-21. doi: 10.1177/1557988314537517. Epub 2014 Jun 4. PMID 24899517
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Daubenmier, J. J. The relationship of yoga, body awareness, and body responsiveness to self-objectification and disordered eating. Psychology of Women Quarterly. 2005; 29(2): 207-219.
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Frayeh, & Lewis, B. A. The effect of mirrors on women's state body image responses to yoga. Psychology of Sport and Exercise. 2018; 35: 47-54.
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Lakens D. Calculating and reporting effect sizes to facilitate cumulative science: a practical primer for t-tests and ANOVAs. Front Psychol. 2013 Nov 26;4:863. doi: 10.3389/fpsyg.2013.00863. PMID 24324449
- [Background] Lindner, D., & Tantleff-Dunn, S. The development and psychometric evaluation of the Self-Objectification Beliefs and Behaviors Scale. Psychology of Women Quarterly. 2017; 41(2): 254-272.
- [Background] Menzel, & Levine, M. P. Embodying experiences and the promotion of positive body image: The example of competitive athletics. In Self-objectification in women: Causes, consequences, and counteractions. Washington, DC: American Psychological Association. 2011; (pp. 163-186).
- [Background] Radloff, L. S. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977; 1(3): 385-401.
- [Background] Reboussin, B. A., Rejeski, W. J., Martin, K. A., Callahan, K., Dunn, A. L., King, A. C., & Sallis, J. F. Correlates of satisfaction with body function and body appearance in middle- and older aged adults: The activity counseling trial (ACT). Psychology & Health. 2000; 15(2): 239-254.
- [Background] Sandoz, E. K., Wilson, K. G., Merwin, R. M., & Kellum, K. K. Assessment of body image flexibility: The body image-acceptance and action questionnaire. Journal of Contextual Behavioral Science. 2013; 2(1-2): 39-48.